CLINICAL TRIAL: NCT04726657
Title: Comparison of Two Biphasic Insulin Regimens in Well-controlled Patients With the Use of Continuous Glucose Monitoring and New Glycemic Control Indices
Brief Title: Comparison of Two Biphasic Insulin Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Triantafyllos Didangelos, Associate Professor of Internal Medicine-Diabetology, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2279
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus type 2; glycemic control; glycated albumin; continuous glucose monitoring; fructosamine; glycated hemoglobin; insulin; premixed human insulin; premixed insulin analog
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Intervention Model Description: Cross-over
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Premixed Insulin (Active Comparator): Premixed Human Insulin
  Interventions: Drug: Premixed Human Isophane Insulin Suspension + Human Insulin Injection; Drug: Premixed Insulin
- Premixed insulin (Active Comparator): Premixed Insulin Analog
  Interventions: Drug: Premixed Human Isophane Insulin Suspension + Human Insulin Injection; Drug: Premixed Insulin

INTERVENTIONS:
Drug: Premixed Human Isophane Insulin Suspension + Human Insulin Injection — premixed human insulin
  Other Names: premixed human insulin
Drug: Premixed Insulin — Premixed Insulin Analog Biphasic Aspart 30
  Other Names: Biphasic Aspart 30

SUMMARY:
Comparison of Two Biphasic Insulin Regimens in Well-controlled Patients With the Use of Continuous Glucose Monitoring and New Glycemic Control Indices

DETAILED DESCRIPTION:
A cross-over study of 36 well controlled people with type 2 Diabetes Mellitus who underwent 7-day Continuous Glucose Monitoring with Premixed Human Insulin 30/70 and subsequently with Biphasic Aspart 30.

ELIGIBILITY:
Inclusion Criteria:

* regular attendees of Outpatient Clinic of the Diabetes Centre of the 1st Department of Internal Medicine of University Hospital in Thessaloniki Greece
* The patients were on Premixed Human Insulin 30/70 twice daily with or without metformin
* baseline HbA1c<7%

Exclusion Criteria:

* the presence of type 1 Diabetes Mellitus
* stage 4 Chronic Kidney Disease
* use of antidiabetic medications other than insulin and metformin
* major cardiovascular event during the last six months
* acute illness and hospitalization during the last two weeks
* pregnancy
* absence of good metabolic control assessed with self-monitoring of blood glucose during the week before entering the study (>20% of the measurements <80mg/dl or >130mg/dl)
* inability of the patients to understand the study procedures and sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Change in average blood glucose | 7 days
  average blood glucose (mg/dl) from continuous glucose monitoring
Glycated Albumin | 7 days
  levels of glycated albumin (%) in serum
Fructosamine | 7 days
  levels of fructosamine (μmol/L) in serum

SECONDARY OUTCOMES:
Daily Insulin requirements | 7 days
  change in total daily dose of insulin (u)
nocturnal average blood glucose | 7 days
  change in nocturnal average blood glucose
Time in range | 7 days
  change in time in range (% and minutes) from continuous glucose monitoring
time above 180 | 7 days
  change in time above 180 (% and minutes) from continuous glucose monitoring
time below 70 | 7 days
  change in time below 70 (% and minutes) from continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Triantafyllos Didangelos, Assoc. Prof., Principal Investigator — AHEPA Hospital Aristotle University Of Thessaloniki

IPD SHARING:
Plan to Share IPD: No
Upon request